CLINICAL TRIAL: NCT05847478
Title: Effects of Auricular Acupressure Versus Intermittent Dietary Restriction in Children With Gastric Heat and Dampness Obstruction: a Randomized Controlled Trial
Brief Title: Effects of Auricular Acupressure Versus Intermittent Dietary Restriction in Children With Gastric Heat and Dampness Obstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AP_IDR_2.0
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Obesity, Childhood
Keywords: Auricular acupressure; Intermittent dietary restriction; Gastric Heat and Dampness Obstruction
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupressure therapy group (AAT) (Experimental): The participants will be randomly assigned to receive the auricular point patch therapy. The intervention period is 3 months.
  Interventions: Other: Auricular acupressure of traditional Chinese Medicine; Behavioral: Health education
- Intermittent low carbohydrate diet group (ILCD) (Experimental): The participants will be randomly assigned to receive the intermittent low carbohydrate diet. The duration of the study is 3 months, including 1-month intervention period and 2-month self maintenance period.
  Interventions: Behavioral: Intermittent low carbohydrate diet; Behavioral: Health education

INTERVENTIONS:
Other: Auricular acupressure of traditional Chinese Medicine — The participants will be randomly assigned to receive the auricular point patch therapy.
  The selected acupoints include Shenmen, hungry point, endocrine, stomach, mouth and subcortical. The opaque patch with vaccaria seed is used for acupoint pressing. Pressing the acupoints once a day before and after eating, each time for 1 minute, lasting for 2-3 days, follow up visit once a week. The intervention period is 3 months.
  Arms: Auricular acupressure therapy group (AAT)
Behavioral: Intermittent low carbohydrate diet — The participants will be randomly assigned to the intermittent low carbohydrate diet group.
  The intermittent carbohydrate diet includes 7 days of low carbohydrate diet within 2 weeks (consecutive or nonconsecutive, carbohydrate intake be controlled as ≤ 50g per day). The study duration is 3 months, including 1-month intervention period and 2-month self-maintenance period.
  Arms: Intermittent low carbohydrate diet group (ILCD)
Behavioral: Health education — Health education is conducted once a week during 3-month intervention for all participants. Health education including the understanding of childhood obesity and cardiovascular disease, how to determine the cardiometabolic risk level, and the lifestyle intervention as caloric restriction and increased physical activity to promote health.

SUMMARY:
This is a three-month randomized controlled trial to investigate the effects of auricular acupressure versus Intermittent carbohydrate restriction on cardiometabolic risk in obese children with gastric heat and dampness obstruction.

DETAILED DESCRIPTION:
Obesity in childhood is associated with multiple cardiometabolic risk factors including hyperglycemia, dyslipidemia and hypertension, which predicts increased risk for developing obesity-driven complications in adulthood. Auricular acupuncture therapy is an intervention with purported success for the treatment of obesity. However, traditional intervention rarely has long-term success in children and adolescents. Low-carbohydrate diets have also been shown to reduce body weight and improve insulin sensitivity in children.

This is a three-month randomized controlled trial in children with gastric damp-heat obstruction, in order to explore the effects of traditional Chinese medicine auricular acupressure and intermittent carbohydrate restriction on cardiovascular metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one of the following cardiometabolic risk factors: overweight or obesity, prediabetes, dyslipidemia or elevated blood pressure.
* Traditional Chinese medical syndrome type is gastric heat and dampness obstruction syndrome.

Exclusion Criteria:

* Diagnosis of obesity associated with genetic or endocrine diseases, including hypercortisolism, polycystic ovary syndrome, primary hypothyroidism and hypothalamic obesity.
* Participating in other clinical trials or have participated in other clinical trials in recent 3 months.
* Diagnosis of organic diseases, including heart, liver, kidney and brain or infectious diseases and mental diseases.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | From baseline to one month after intervention
  The body weight will be measured by fixed research staff at baseline and one month after intervention.

SECONDARY OUTCOMES:
changes in the cumulative score of traditional Chinese medicine syndromes | From baseline to three month after intervention
  The investigators will measure the change in scores of chinese medicine symptoms according to the Traditional Chinese Medicine Guideline Scale: 0 - 3. 0 = None. 1 = Mild. 2 = Moderate. 3= Severe
Changes in glucose metabolism level, including fasting blood glucose, glycated hemoglobin, insulin level, etc | From baseline to three month after intervention
  Serum from fasting blood sample is used for measurement of glucose metabolism at baseline, one month and three month after intervention.
Changes in waist-to-height ratio(WtHR), body mass index (BMI) and blood pressure | From baseline to three month after intervention
  The weight、height、waist circumference and blood pressure will be measured by fixed research staff at baseline , one month and three month after intervention. BMI and WtHR are calculated using the corresponding equation.
Changes in body fat content | From baseline to three month after intervention
  Body composition involves measuring the body fat percentage by using the LUNAR DPX Dual Energy X-ray Absorptiometry (DXA) equipment (General Electric Company, USA)) at baseline , one month and three month after intervention.
Changes in blood lipid ,liver and kidney function level | From baseline to three month after intervention
  Serum from fasting blood sample is used for measurement of blood lipid ,liver and kidney function at baseline, one month and three month after intervention.
Changes in Gut microbiota | From baseline to one month after intervention
  Stool samples are collected with Boyou®- nucleic acid storage tube and stored in the laboratory -80℃ refrigerator at the baseline and one month after intervention. For the study of intestinal flora diversity, the 16SrDNA target region is amplified, and the information of intestinal microbial diversity and community composition is obtained by detecting the sequence variation and abundance of the target region.
Changes in dietary and exercise data | From baseline to three month after intervention
  Diet and exercise data are recorded by the children and their families, but they will be educated by qualified clinicians before recording.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

REFERENCES:
- [Derived] Sun W, He J, Wang W, Lu C, Lin Y, Dou Y, Yan W, Yu J. Auricular Acupressure Versus an Intermittent Low-Carbohydrate Diet in Children With Overweight or Obesity With Gastric-Heat and Dampness-Obstruction Syndrome: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 3;14:e59856. doi: 10.2196/59856. PMID 40053799